CLINICAL TRIAL: NCT02264691
Title: UTMB Research on Severe Asthma (UROSA) Study
Acronym: UROSA
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 08-128
Record Dates: First submitted 2014-10-08; First posted 2014-10-15 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Normal (healthy volunteers): No Research Intervention. Clinically indicated interventions only.
- Mild Asthmatics: No Research Intervention. Clinically indicated interventions only.
- Mild to Moderate Asthmatics: No Research Intervention. Clinically indicated interventions only.
- Severe Asthmatics: No Research Intervention. Clinically indicated interventions only.

SUMMARY:
To identify and understand biologic aspects of severe asthma compared to subjects with mild to moderate asthma and subjects without asthma (normal or healthy volunteers).

DETAILED DESCRIPTION:
It has been shown that severe asthma differs from milder asthma in its pathophysiology; in particular we are interested in examining why patients with severe asthma have disease that is resistant to corticosteroids. While we will be studying patients with severe asthma, we also need to study subjects to act as controls. To this end we will recruit subjects into the following groups: Normal volunteers; Mild asthmatics not taking inhaled corticosteroids; Mild to moderate asthmatics requiring and using inhaled corticosteroids and Severe asthmatics.

Subjects between the ages of 18 and 65 will be enrolled in this study. We aim to recruit enough subjects such that 120 male and female participants (30 in each of the above groups) will complete the bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be in good general health (with exception to asthma). • Normal controls / healthy volunteers (NC) subjects with no past history of asthma or other lung disease. To determine this, subjects must have an FEV1 equal to or greater than 80% of predicted value and have a normal FEV1/FVC ratio.

Asthma subjects Eligible asthmatic participants must have a physician diagnosis of asthma for at least 1 year. Participants must either have historical evidence of reversibility of FEV1 of at least 12%, or demonstrate such a change during the study visits, or must have historical evidence of a PC20 for methacholine < 8mg/ml.

* Mild Asthma with no Corticosteroids (MANC) will be defined as control of asthma with short acting β2-agonists or leukotrine antagonist or both, but not requiring inhaled corticosteroids.
* Mild to Moderate asthma (MMA) will be defined as control of asthma with an inhaled corticosteroid (less than or equal to 250 mcg daily inhaled fluticasone equivalent) in addition to the medications listed in the MANC group or long acting β2-agonists.
* Severe asthma (SA) will be defined according to the ATS criteria for Refractory Asthma (10)

Exclusion Criteria:

* Exclusion criteria apply for all subjects:

  * Current smoker, or former smoker with >10 pack years history or having quit within the past year
  * Asthma exacerbation, requiring a new or increased dose of oral corticosteroids, within the past 30 days
  * Pregnant or lactating female
  * Significant/uncontrolled medical condition (uncontrolled diabetes, coronary artery disease, uncontrolled hypertension)
  * Diagnosis of emphysema or other significant pulmonary disease
  * If, in the opinion of the PI (WJC) the subject has co-morbid conditions that make them unsafe to undergo bronchoscopy, subjects will be given the choice to withdraw from the study or allowed to complete visits 1-3 only.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal volunteers; Mild asthmatics not taking inhaled corticosteroids; Mild to moderate asthmatics requiring and using inhaled corticosteroids and Severe asthmatics
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2009-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
evaluate patients with severe asthma | 7 Years
  To evaluate patients with severe asthma and to establish the mechanisms by which the lack of response to treatment may occur.

CONTACTS AND LOCATIONS:
Overall Officials: William Calhoun, M.D., Principal Investigator — UTMB
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States